CLINICAL TRIAL: NCT02297620
Title: Specified Drug Use resulTs survEy of IpragLifLozin treAtment in ELDERly type2 Diabetes Patients (STELLA-ELDER)
Brief Title: The Survey of Ipragliflozin Treatment in Elderly type2 Diabetes Patients
Acronym: STELLA-ELDER
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SGL001
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes
Keywords: SGLT-2 inhibitor; Elderly patients; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suglat group
  Interventions: Drug: Suglat®

INTERVENTIONS:
Drug: Suglat® — oral
  Other Names: ipragliflozin

SUMMARY:
The objective of this survey is to confirm the safety of Suglat Tablets when used in the elderly.

DETAILED DESCRIPTION:
Elderly patients (65 years or older at the time of first administration) with type 2 diabetes who used Suglat Tablets within 3 months from its launch are included in this study. Followings are measured with the patients.

1. Specify incidence rates of adverse drug reactions associated with a decrease in body fluids and their risk factors.
2. Investigate the occurrence of urinary tract infection.
3. Investigate the occurrence of adverse drug reactions in patients at a high risk (those who have poorly controlled blood sugar levels, concurrent organic abnormalities in the urinary system, advanced diabetic neuropathy, etc).
4. Investigate the occurrence of adverse drug reactions other than the above.
5. Factors that may possibly influence the safety of Suglat Tablets.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes who used Suglat Tablets within 3 months from its launch

Exclusion Criteria:

* off-label use patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with type 2 diabetes who used Suglat Tablets within 3 months from its launch
Sampling Method: Non-Probability Sample
Enrollment: 8687 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Specify incidence rates of adverse drug reactions associated with a decrease in body fluids and their risk factors | Up to 12 months

SECONDARY OUTCOMES:
Investigate the occurrence of urinary tract infection | 1-month, 3-month, 6-month, 9-month and 12-month (or at treatment discontinuation time)
Investigate the occurrence of adverse drug reactions in patients at a high risk (those who have poorly controlled blood sugar levels, concurrent organic abnormalities in the urinary system, advanced diabetic neuropathy, etc). | 1-month, 3-month, 6-month, 9-month and 12-month (or at treatment discontinuation time)
Investigate the occurrence of adverse drug reactions other than the above | 1-month, 3-month, 6-month, 9-month and 12-month (or at treatment discontinuation time)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shikoku
  - Tōhoku

REFERENCES:
- [Derived] Terauchi Y, Yokote K, Nakamura I, Sugamori H. Safety of ipragliflozin in elderly Japanese patients with type 2 diabetes mellitus (STELLA-ELDER): Interim results of a post-marketing surveillance study. Expert Opin Pharmacother. 2016;17(4):463-71. doi: 10.1517/14656566.2016.1145668. Epub 2016 Feb 5. PMID 26800061